CLINICAL TRIAL: NCT03901066
Title: Smoking Dependence (Fagerström) as a Relevant Indicator for Tobacco Related Studies in Periodontology.
Brief Title: Smoking Dependence and Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Leila Salhi, periodontist, PhD student, University of Liege
Other Study IDs: File number: B707201419816
Record Dates: First submitted 2019-03-22; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Smoking; Periodontitis
MeSH Terms: conditions — Smoking; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study was designed as a, single-center, prospective cohort study focusing on the relationship between smoking status and the severity of periodontitis

DETAILED DESCRIPTION:
The present study was designed as a, single-center, prospective cohort study focusing on the relationship between smoking status and the severity of periodontitis.

The research question was " How the Fagerström for nicotine dependence (FTND) and the number of cigarette cunsuption (NNC) are correlated to the severity of chronic periodontitis"? Thirty-four consecutive smoker patients presenting a chronic periodontitis were included in the study, and the smoking status was defined both by NCC and FTND.

Periodontal clinical parameters were correlated with NCC and FTND.

All the clinical periodontal parameters were recorded by a single periodontist (L.S). Periodontal assessments included: probing depth (PD), gingival recession (RD), clinical attachment level (CAL), bleeding on probing (BOP), plaque score index (PI), Furcation (Furc), tooth mobility and the percentage of sites of PD ≥ 6mm. A graduated manual periodontal probe was used to take measurements at the 6 sites of each tooth. BOP (%) and plaque score (%).

All the participants of the study respected the following inclusion criteria: 1/ smoker patients aged of minimum 18 years old, 2/ chronic periodontitis, 3/ presence of a minimum of 6 teeth at each arch, 4/ a minimum of 6 teeth with pocket depth of 5 mm, 5/ signed the informed consent. The exclusion criteria were: 1/ aggressive periodontitis, 2/ diabetes, 3/ connective tissue disease, 4/ pregnancy, 5/ radio-therapy, 6/ chemotherapy, 7/ psychological disease, 8/ previous periodontal therapy.

The patient smoking status was defined by FTND and NCC FTND scores were categorized in 3 groups

* scores < 4 for low nicotine dependence,
* scores = 4-5 for moderate nicotine dependence
* scores > 5 for high nicotine dependence.

The NCC s was classified in three levels of smokers as described in most of the periodontal studies:

* Number of cigarette smoking ≤ 10 per day for low consumption
* Number of cigarette smoking from 10 to 20 per day for moderate consumption
* Number of cigarette smoking > 20 per day for high cigarette consumption

ELIGIBILITY:
Inclusion Criteria:

* smoker patients aged of minimum 18 years old
* chronic periodontitis
* presence of a minimum of 6 teeth at each arch
* a minimum of 6 teeth with pocket depth of 5 mm
* signed the informed consent

Exclusion Criteria:

* aggressive periodontitis
* diabetes
* connective tissue disease
* pregnancy
* radio-therapy
* chemotherapy
* psychological disease
* previous periodontal therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 34 consecutive smoker patients presenting periodontitis were included from the Department of Periodontology and Oral Surgery at the University of Liege, Belgium. All the participants of the study respected the aboveinclusion criteria
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
effect of nicotine dependence level on periodontal outcomes | 1 day
  effect of nicotine dependence score on pocket depth (PD)